CLINICAL TRIAL: NCT01566162
Title: A Twelve Week, Multicenter, Open Label Extension Study in Subjects With Schizophrenia
Brief Title: A Twelve Week, Open Label Extension Study in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1050307; 2011-004790-90 (EudraCT Number)
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Results first posted 2014-11-20 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Schizophrenia
Keywords: Lurasidone; Latuda; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lurasidone (Experimental): Lurasidone 40 - 80mg flexible dose
  Interventions: Drug: Lurasidone

INTERVENTIONS:
Drug: Lurasidone — Lurasidone 40-80 mg taken orally taken once daily

SUMMARY:
This is a 12-week, multi-center, open-label extension study designed to evaluate the longer-term safety, tolerability and effectiveness of lurasidone for the treatment of subjects with schizophrenia.

DETAILED DESCRIPTION:
This is a 12-week, multi-center, open-label extension study designed to evaluate the longer-term safety, tolerability and effectiveness of lurasidone for the treatment of subjects with schizophrenia who have participated in Study D1050238, a double-blind, placebo-controlled, randomized withdrawal study of lurasidone for the maintenance treatment of subjects with schizophrenia. Subjects who have completed the 28-week double-blind phase or who have experienced a protocol-defined relapse event during the double-blind phase of study D1050238 will have the option to participate in this study. In addition, if/when the study is discontinued by the sponsor, all subjects participating in the open-label phase and the double-blind phase of study D1050238 will have the option to participate in this extension study

ELIGIBILITY:
Inclusion Criteria:

* Subject has agreed to participate by providing written informed consent.
* Subject will be eligible to participate if one of the following criteria is met:
* Subject has completed the 28-week double-blind phase of study D1050238
* Subject has experienced a protocol-defined relapse event during the double- blind phase in study D1050238
* Subject is participating in the open-label or double-blind phase of study D1050238 if/when study D1050238 is terminated by the sponsor.
* Subject has completed all required assessments on the final study visit (Study Visit Number 42) in study D1050238.
* Subject is judged by the Investigator to be suitable for participation in a 12-week clinical trial involving open-label lurasidone treatment and is able to comply with the protocol in the opinion of the Investigator.

Exclusion Criteria:

* Subject is considered by the investigator to be at imminent risk of suicide or injury to self, others, or property.
* Subject answers "yes" to "Suicidal Ideation" item 4 (active suicidal ideation with some intent to act, without specific plan) or item 5 (active suicidal ideation with specific plan and intent) on the C-SSRS at the extension baseline visit (Study Visit Number 42 in study D1050238). Subjects who answer "yes" to this question must be referred by the Investigator for appropriate follow-up evaluation and treatment.
* Subject tests positive for drugs of abuse or is suspected of current alcohol abuse at the extension baseline visit (Study Visit Number 42 in study D1050238). In the event a subject tests positive for cannabinoids, the Investigator will evaluate the subject's ability to abstain from cannabis during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2012-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lurasidone Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (63):
- United States (38):
  - K and S Professional Research Services, Little Rock, Arkansas
  - Woodland International Research Inc., Little Rock, Arkansas
  - Comprehensive Clinical Development Inc., Cerritos, California
  - Diligent Clinical Trials, Downey, California
  - Synergy Clinical Research Center, Escondido, California
  - CNS Network, Garden Grove, California
  - AXIS Clinical Trials, Los Angeles, California
  - Synergy Clinical Research Center, National City, California
  - Excell Research, Inc., Oceanside, California
  - CNRI-Los Angeles. LLC, Pico Rivera, California
  - California Neuropsychopharmacolgoy Clinical Research Insitute, San Diego, California
  - Neuropsychiatric Research Center of Orange County, Santa Ana, California
  - Collaborative Neuroscience Network, Torrance, California
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Accurate Clinical Trials, Kissimmee, Florida
  - Galiz Research, Miami Springs, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Comprehensive NeuroScience Inc., Atlanta, Georgia
  - Lake Charles Clinical Trials, LLC, Lake Charles, Louisiana
  - Lousiana Clinical Research, LLC, Shreveport, Louisiana
  - Center for Behavioral Health, LLC, Rockville, Maryland
  - Psychiatric Care and Research Center, O'Fallon, Missouri
  - Psych Care Consultants Research, St Louis, Missouri
  - Robert Lynn Horne, MD, Las Vegas, Nevada
  - CRI Worldwide LLC, Willingboro, New Jersey
  - Erie County Medical Center, Corp, Buffalo, New York
  - Neurobehavioral Research Inc., Cedarhurst, New York
  - Comprehensive Clinical Development, Inc, Fresh Meadows, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Oklahoma Clinical Research, Oklahoma City, Oklahoma
  - CRI Worldwide LLC at Kirkbride, Philadelphia, Pennsylvania
  - Lincoln Research, Lincoln, Rhode Island
  - Community Clinical Research, Inc., Austin, Texas
  - FutureSearch Clinical Trials LP, Austin, Texas
  - FutureSearch Clinical Trials, LP, Dallas, Texas
  - Pillar Clinical Research, LLC, Dallas, Texas
  - Department of Psychiatry, University of Utah Health Sciences Center, Salt Lake City, Utah
- France (2):
  - Centre Hospitalier Spécialisé (CHS) du Jura - Centre Médico Psychiatrique (CMP), Dole
  - Hôpital Chalucet, Centre hospitalier intercommunal de Toulon la Seyne sur mer (CHITS), Toulon
- Italy (2):
  - Dipartimento Salute Mentale ASL 1, Massa
  - A.O.U. Santa Chiara, U.O di Psichiatria 1 building n.4, Pisa
- Russia (6):
  - Regional Government Institution (RGI) 'Lipetsk Regional Psychoneurology Hospital', Lipetsk
  - Limited Liability Company (LLC) 'Research Center For Treatment and rehabilitation 'Phoenix', Rostov-on-Don
  - St. Petersburg State Healthcare Institution (SPbSHI) "City Psychiatric Hospital #6", Saint Peterburg
  - St. Petersburg State Budgetary Healthcare Institution 'City Psychoneurology Dispensary #7 (with In-Patient Department)', (SPb SBHI "CPNDD-7"), Saint Petersburg
  - St. Petersburg State Budgetary Healthcare Institution 'City Psychoneurology Dispensary #7 (with In-Patient Department)', (SPb SBHI "CPNDD-7"), at Daycare Facility #1, Saint Petersburg
  - St. Petersburg State Government Healthcare Institution "City Psychiatric Hospital #4" (St. Petersburg Insane Asylum Distributor), Saint Petersburg
- Serbia (6):
  - Military Medical Academy, Clnic for Psychiatry, Belgrade
  - Institute of Mental Health, Dusica
  - Clinical Centre Kragujevac, Clinic for psychiatry, Kragujevac
  - Clinical Centre Nis, Clinic for mental health protection, Niš
  - Specialized hospital for psychiatric diseases "Sveti Vracevi", Novi Kneževac
  - Clinical Centre Vojvodine, Clinic for Psychiatry, Novi Sad
- Slovakia (6):
  - Nemocnica s poliklinikou v Prievidzi so sidlom v Bojniciach, Psychiatricke oddelenie, Bojnice
  - Psychiatricka ambulancia Mentum s.r.o., Bratislava
  - Psychiatricka nemocnica Michalovce n.o., Michalovce
  - PsychoLine s.r.o. Psychiatricka ambulancia, Rimavská Sobota
  - Nemocnica s poliklinikou sv Barbory Roznava a.s. Psychiatricke oddelenie, Rožňava
  - "Centrum zdravia R.B.K., spol. s.r.o., Svidník
- South Africa (3):
  - Cape Trial Centre, Tygervalley, Western Cape
  - Research Unit, Department of Psychiatry Free State Psychiatric Complex, Bloemfontein
  - Denmar Hospital Consulting Rooms, Pretoria

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lurasidone
Started | 191
Completed | 155
Not Completed | 36

BASELINE CHARACTERISTICS:
Arm/Group | Lurasidone
Number analyzed (Participants) | 191
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.7 (12.30)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 190
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76
  Male | 115
Region of Enrollment [Number; unit: participants]
  Serbia | 22
  France | 4
  United States | 114
  Slovakia | 15
  Russia | 19
  South Africa | 17

OUTCOME MEASURES:

1. Primary Outcome: Safety - Treatment-emergent Adverse Events (TEAEs), TEAEs Leading to Discontinuation, and Serious AEs (SAEs)
Description: Number of subjects with treatment-emergent adverse events (TEAEs), TEAEs leading to discontinuation, and serious AEs (SAEs)
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Lurasidone
Number analyzed (Participants) | 191
participants
  Subjects with TEAEs | 72
  TEASs leading to discontinuation | 7
  Subjects with TESAEs | 13

2. Primary Outcome: Efficacy - Change in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: The PANSS is an interview-based measure of the severity of psychopathology in adults with psychotic disorders. The measure is comprised of 30 items. An anchored Likert scale from 1-7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. The PANSS total score is the sum of all 30 items and ranges from 30 through 210. A higher score is associated with greater illness severity.
Time Frame: Baseline to week 12 LOCF endpoint
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone
Number analyzed (Participants) | 191
units on a scale | -8.4 (15.06)

3. Primary Outcome: Efficacy - Change From Baseline in Clinical Global Impression-Severity of Illness (CGI-S) Score.
Description: The CGI-S score is a single value, clinician-rated assessment of illness severity and ranges from 1= 'Normal, not at all ill' to 7= 'Among the most extremely ill patients'. A higher score is associated with greater illness severity.
Time Frame: Baseline to week 12 LOCF endpoint
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone
Number analyzed (Participants) | 191
units on a scale | -0.48 (1.051)

4. Secondary Outcome: Change From Baseline in Montgomery -Asberg Depression Rating Scale Total Score
Description: The MADRS consists of 10 items, each rated on a Likert scale, from 0="Normal" to 6="Most Severe". The MADRS total score is calculated as the sum of the 10 items. The MADRS total score ranges from 0 to 60. Higher scores are associated with greater severity.
Time Frame: Baseline to week 12 LOCF endpoint
Population: Only 182 subjects had post-baseline MADRS assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone
Number analyzed (Participants) | 182
units on a scale | -3.3 (7.83)

5. Secondary Outcome: Short Form-12 Health Survey (SF-12)
Description: The SF-12v2 is a self-administered, multipurpose short-form (SF) generic measure of health status. It was developed to be a shorter, yet valid, alternative to the SF-36 for use in large surveys of general and specific populations as well as in large longitudinal studies of health outcomes. The 12 items in the SF-12v2 are a subset of those in the SF-36; SF-12v2 includes one or two items from each of the eight health concepts with higher scores indicative of higher functioning and better health. The Physical Component Score is a composite of the Physical Functioning, Role Functioning, Bodily Pain and General Health scales. Physical Composite Scores (PCS) is computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Time Frame: Baseline to week 12 LOCF endpoint
Population: Only 182 subjects had post-baseline SF-12.v2 assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone
Number analyzed (Participants) | 182
units on a scale | -0.45 (6.642)

6. Secondary Outcome: Modified Specific Levels of Functioning (SLOF) Total Score.
Description: The modified SLOF scale is designed to measure directly observable behavioral functioning and daily living skills of patients with chronic mental illness. The modified SLOF consists of 24 items, each item is rated on a 5-point scale and mapped to 0 to 4. The total score will be the sum of all 24 items and ranges from 0 to 96. A higher score indicates worse condition.
Time Frame: 12 weeks
Population: Only 174 subjects had SLOF assessments at week 12 LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone
Number analyzed (Participants) | 174
units on a scale | -1.8 (9.55)

7. Secondary Outcome: Brief Adherence Rating Scale (BARS)
Description: The Brief Adherence Rating Scale (BARS) is a clinician-administered adherence assessment instrument that consists of four items including three questions and a visual analog rating scale (VAS) to assess the percentage (0 100%) of doses taken by the subject in the previous month.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of monthly doses taken
Arm/Group | Lurasidone
Number analyzed (Participants) | 182
percentage of monthly doses taken | 99.0 (3.08)

8. Secondary Outcome: Smoking Questionnaire
Description: Smoking questionnaire - average number of cigarettes per day at week 12 (LOCF).
Time Frame: 12 weeks
Population: Only 36 subjects who were smokers had the smoker questionnaire assessments.
Measure: Mean (Standard Deviation); unit: number of cigarettes smoked daily
Arm/Group | Lurasidone
Number analyzed (Participants) | 36
number of cigarettes smoked daily | 11.1 (9.95)

9. Secondary Outcome: Intent to Attend Assessment
Description: The ITA assessment will be administered by a research staff member. The response is recorded on a 10-point scale, with 0 = "Not at all" and 9 = "Extremely". The ITA allowed the site to capture data regarding dropout risk. The following question was completed at the baseline visit: "How likely is it that you will complete the study?"
Time Frame: 12 weeks
Population: Only 1825 subjects answered the questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone
Number analyzed (Participants) | 185
units on a scale | 8.3 (1.14)

ADVERSE EVENTS:
Time Frame: 12 Weeks
Arm/Group | Lurasidone
Serious Adverse Events (participants affected / at risk) | 13/191
Other Adverse Events (participants affected / at risk) | 34/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone (N=191)
Artrial flutter (Cardiac disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Schizophrenia (Psychiatric disorders) | 6 (6)
Psychotic Disorder (Psychiatric disorders) | 4 (5)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone (N=191)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (5)
Nasopharyngitis (Infections and infestations) | 5 (5)
Akathisia (Nervous system disorders) | 10 (10)
Headache (Nervous system disorders) | 4 (5)
Schizophrenia (Psychiatric disorders) | 8 (8)
Anxiety (Psychiatric disorders) | 4 (9)
Insomnia (Psychiatric disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS agreement between Principal Investigator and Sponsor that restricts PI's rights to discuss or publish trial results after trial is completed.

In addition to the <60-180 day restriction above, since this is a multicenter study, 1st publication of study results shall be made with other participating study sites as a multicenter publication provided, if a multicenter publication is not forthcoming within 24 months post completion of study at all sites, PI shall be free to publish.